CLINICAL TRIAL: NCT05621915
Title: Nadroparin Pharmacokinetics in Different Stages of COVID-19-a Prospective Observational Study.
Brief Title: Nadroparin Pharmacokinetics in Different Stages of COVID-19
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Collaborators: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Paweł Piwowarczyk, Principal Investigator, Medical University of Lublin
Other Study IDs: KE 0254/23/2021
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Thrombosis; Nadroparin; COVID-19; Mechanical Ventilation; Anticoagulants and Bleeding Disorders
MeSH Terms: conditions — Thrombosis; COVID-19; Hemostatic Disorders | interventions — Nadroparin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- conventional oxygen therapy: Patients treated with conventional oxygen in Infectious Diseases Ward.
  Interventions: Drug: Nadroparin
- mechanical ventilation: Patients who are mechanically ventilated and treated in ICU.
  Interventions: Drug: Nadroparin
- mechanical ventilation and ECMO: Patients who are mechanically ventilated and on ECMO treated in ICU.
  Interventions: Drug: Nadroparin

INTERVENTIONS:
Drug: Nadroparin — Subcutaneous injection of nadroparin according to the ICU guidelines for thromboprophylaxis in ICU patients.

SUMMARY:
Objective:

The risk of thrombotic complications in critical COVID-19 patients remains extremely high, and multicenter trials failed to prove the survival benefit of escalated doses of low molecular weight heparins (LMWH) in this group. The aim of this study was to develop a pharmacokinetic model of LMWH (nadroparin calcium) according to different stages of COVID-19 severity.

Design:

The investigators performed a prospective observational study.

Patients:

Blood samples were obtained from 43 COVID-19 patients that received nadroparin and were treated with conventional oxygen therapy, mechanical ventilation, and extracorporeal membrane oxygenation.

Setting:

The investigators recorded clinical, biochemical, and hemodynamic variables during 72 hours of treatment. The analyzed data comprised 782 serum nadroparin concentrations and 219 anti-factor Xa levels. The investigators conducted population nonlinear mixed-effects modeling (NONMEM) and performed Monte Carlo simulations of the probability of target attainment (PTA) for reaching 0.2-0.5 IU/ml anti-Xa levels in study groups.

Interventions: None.

Measurements and Main Results:

The investigators successfully developed a one-compartment model to describe the population pharmacokinetics of nadroparin in different stages of COVID-19.

Conclusions:

Different nadroparin dosing is required for patients undergoing mechanical ventilation and ECMO to achieve the same targets as those for non-critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in the Department of Anesthesiology and Intensive Care and the Department of Infectious Diseases of a tertiary academic hospital with confirmed SARS-CoV-2 infection with a real-time reverse transcription polymerase chain reaction (RT-PCR) or an antigen test.

Exclusion Criteria:

* Coagulation disorders at the start of the therapy.

Age Groups: Child, Adult, Older Adult
Study Population: First group (Group 1) consisted of 14 patients treated with conventional oxygen therapy only in the infectious diseases department. The second group (Group 2) consisted of 14 mechanically ventilated patients treated in the ICU, and the third group (Group 3) was formed by 15 patients supported with extracorporeal membrane oxygenation (ECMO) and mechanically ventilated in the ICU. The investigators used surviving sepsis campaign guidelines for COVID-19 for the escalation of treatment in the study population.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Change in nadroparin concentration in blood measurement | 6 hours
  Sequential measurement every 6 hours
Change in anti-Xa serum level | 12 hours
  Sequential measurement every 12 hours

SECONDARY OUTCOMES:
Volume of distribution of nadroparin | 24 hours
Clearance of nadroparin | 24 hours
Absorption rate of nadroparin | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Piwowarczyk, MD PhD, Principal Investigator — Medical University of Lublin
Locations (1):
- 2nd Department of Anesthesiology and Critical Care, Medical University of Lublin, Lublin, Lublin Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Piwowarczyk P, Szczukocka M, Cios W, Okunska P, Raszewski G, Borys M, Wiczling P, Czuczwar M. Population Pharmacokinetics and Probability of Target Attainment Analysis of Nadroparin in Different Stages of COVID-19. Clin Pharmacokinet. 2023 Jun;62(6):835-847. doi: 10.1007/s40262-023-01244-4. Epub 2023 Apr 25. PMID 37097604